CLINICAL TRIAL: NCT02031666
Title: A Single-Dose, Open-Label, Randomized, Parallel-Group Study to Assess the Relative Bioavailability of 7 Test Tablet Formulations of JNJ-56021927 With Respect to the Capsule Formulation of JNJ-56021927 Under Fasted Conditions in Healthy Male Subjects
Brief Title: A Study to Assess the Relative Bioavailability of 7 Test Tablet Formulations of JNJ-56021927 With Respect to the Capsule Formulation of JNJ-56021927 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aragon Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR103299; 56021927PCR1007 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-10

CONDITIONS: Healthy
Keywords: Healthy; JNJ-56021927; ARN-509; Bioavailability
MeSH Terms: interventions — apalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Treatment A (Active Comparator): 15 participants will receive 240-mg dose as Softgel Capsule Formulation of JNJ-56021927.
  Interventions: Drug: JNJ-56021927 capsule
- Treatment B (Experimental): 15 participants will receive 240-mg dose as Tablet Formulation number 1 of JNJ-56021927.
  Interventions: Drug: JNJ-56021927 tablet
- Treatment C (Experimental): 15 participants will receive 240-mg dose as Tablet Formulation number 2 of JNJ-56021927.
  Interventions: Drug: JNJ-56021927 tablet
- Treatment D (Experimental): 15 participants will receive 240-mg dose as Tablet Formulation number 3 of JNJ-56021927.
  Interventions: Drug: JNJ-56021927 tablet
- Treatment E (Experimental): 15 participants will receive 240-mg dose as Tablet Formulation number 4 of JNJ-56021927.
  Interventions: Drug: JNJ-56021927 tablet
- Treatment F (Experimental): 15 participants will receive 240-mg dose as Tablet Formulation number 5 of JNJ-56021927.
  Interventions: Drug: JNJ-56021927 tablet
- Treatment G (Experimental): 15 participants will receive 240-mg dose as Tablet Formulation number 6 of JNJ-56021927.
  Interventions: Drug: JNJ-56021927 tablet
- Treatment H (Experimental): 15 participants will receive 240-mg dose as Tablet Formulation number 7 of JNJ-56021927.
  Interventions: Drug: JNJ-56021927 tablet

INTERVENTIONS:
Drug: JNJ-56021927 capsule — Participants will receive oral soft gel capsules providing a total dose of 240 mg JNJ-56021927 on Day 1.
  Other Names: ARN-509
  Arms: Treatment A
Drug: JNJ-56021927 tablet — Participants will receive oral tablets providing a total dose of 240 mg JNJ-56021927 on Day 1.
  Arms: Treatment B; Treatment C; Treatment D; Treatment E; Treatment F; Treatment G; Treatment H

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (what the body does to the medication) and relative bioavailability (the extent to which a medication or other substance becomes available to the body) of JNJ-56021927 when administered as 7 test tablet formulations of JNJ-56021927 compared with the softgel capsule formulation of JNJ-56021927 in healthy male participants under fasted conditions at a single dose of 240 mg.

DETAILED DESCRIPTION:
This is a randomized (the study medication is assigned by chance), open-label (all people know the identity of the intervention), single-center, 8-treatment, parallel-group (each group of participants will be treated at the same time) study. Approximately 120 participants (15 participants in each treatment group) will participate in this study. All participants will be randomly assigned to 1 of 8 possible treatments (A, B, C, D, E, F, G, and H). The study will consist of a screening phase (within 21 days before the first administration of the study medication), a treatment phase with 8 parallel single-dose treatments (8 days); a follow up phase (42 days) and an end-of-study or early withdrawal assessments (Day 57). Safety will be evaluated by the assessment of adverse events, clinical laboratory tests, vital signs, and physical examination which will be monitored throughout the study. The duration of participation in the study for an individual participant will be approximately 78 days.

ELIGIBILITY:
Inclusion Criteria:

* During the study and for 3 months after receiving study medication, must agree to use an adequate contraception method (eg, vasectomy, double-barrier, partner using effective contraception), always use a condom during sexual intercourse and to not donate sperm
* Body mass index (weight [kg]/height [m]2) between 18 and 30 kg/m2 and body weight not less than 50 kg
* Blood pressure (after the participant is supine for 5 minutes) between 90 and 140 mmHg systolic, inclusive, and no higher than 90 mmHg diastolic
* A 12-lead electrocardiogram (ECG) consistent with normal cardiac conduction and function
* Non-smoker for 2 months prior to study participation

Exclusion Criteria:

* History of or current clinically significant medical illness including cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders, lipid abnormalities, significant pulmonary disease (including bronchospastic respiratory disease), diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease, and infection
* Clinically significant abnormal values for hematology, clinical chemistry or urinalysis, physical examination, vital signs or 12-lead ECG at screening or at admission to the study center as deemed appropriate by the investigator
* Presence of sexual dysfunction (eg, abnormal libido or erectile dysfunction) or any medical condition that would affect sexual function
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for acetaminophen within 14 days before the first dose of the study drug is scheduled
* History of clinically significant allergies or known hypersensitivity to vitamin E

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2013-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of JNJ-56021927 | Pre-dose, and post-dose Day 1 (0.5, 1, 1.5, 2, 4, 6, 8, 12, 24 hours), Day 2, 3, 4, 5, 6, 7, 8, 15, 22, 29, 36, 43, 50, 57
  The Plasma Concentration (Cmax) is defined as maximum observed analyte concentration.
Time to Reach Maximum Observed Plasma Concentration (Tmax) of JNJ-56021927 | Pre-dose, and post-dose Day 1 (0.5, 1, 1.5, 2, 4, 6, 8, 12, 24 hours), Day 2, 3, 4, 5, 6, 7, 8, 15, 22, 29, 36, 43, 50, 57
  Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Area Under the Plasma Concentration-Time Curve From Time of Administration to 72 hours After Dosing (AUC 0-72h) of JNJ-56021927 | Pre-dose, and post-dose Day 1 (0.5, 1, 1.5, 2, 4, 6, 8, 12, 24 hours), Day 2, 3, 4, 5, 6, 7, 8, 15, 22, 29, 36, 43, 50, 57
  The AUC 0-72h is a measure of the plasma concentration of the drug over time. It is used to characterize drug absorption.
Area Under the Plasma Concentration-Time Curve From Time of Administration to 168 hours After Dosing (AUC 0-168h) of JNJ-56021927 | Pre-dose, and post-dose Day 1 (0.5, 1, 1.5, 2, 4, 6, 8, 12, 24 hours), Day 2, 3, 4, 5, 6, 7, 8, 15, 22, 29, 36, 43, 50, 57
  The AUC 0-168h is a measure of the plasma concentration of the drug over time. It is used to characterize drug absorption.
Area Under the Plasma Concentration-Time Curve From Time Zero to Time at Last Observed Quantifiable Concentration (AUClast) of JNJ-56021927 | Pre-dose, and post-dose Day 1 (0.5, 1, 1.5, 2, 4, 6, 8, 12, 24 hours), Day 2, 3, 4, 5, 6, 7, 8, 15, 22, 29, 36, 43, 50, 57
  The AUClast is area under the plasma concentration-time curve from time zero to the last quantifiable concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) of JNJ-56021927 | Pre-dose, and post-dose Day 1 (0.5, 1, 1.5, 2, 4, 6, 8, 12, 24 hours), Day 2, 3, 4, 5, 6, 7, 8, 15, 22, 29, 36, 43, 50, 57
  The AUC(0-infinity) is area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of Area under Curve (AUC) last and C(last)/lambda(z), in which C(last) is the last observed quantifiable concentration and lambda[z] is the terminal rate-constant of the semi logarithmic drug concentration-time curve.
Elimination Half-Life Period (T1/2) of JNJ-56021927 | Pre-dose, and post-dose Day 1 (0.5, 1, 1.5, 2, 4, 6, 8, 12, 24 hours), Day 2, 3, 4, 5, 6, 7, 8, 15, 22, 29, 36, 43, 50, 57
  The Elimination Half-Life Period (T1/2) is the time measured for the plasma concentration to decrease by 1 half of its original concentration. It is associated with the terminal rate-constant (lambda[z]) of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
First-order Rate Constant of JNJ-56021927 | Pre-dose, and post-dose Day 1 (0.5, 1, 1.5, 2, 4, 6, 8, 12, 24 hours), Day 2, 3, 4, 5, 6, 7, 8, 15, 22, 29, 36, 43, 50, 57
  The first-order rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Time to Last Quantifiable Plasma Concentration (tlast) of JNJ-56021927 | Pre-dose, and post-dose Day 1 (0.5, 1, 1.5, 2, 4, 6, 8, 12, 24 hours), Day 2, 3, 4, 5, 6, 7, 8, 15, 22, 29, 36, 43, 50, 57
Relative Bioavailability (Frel) of JNJ-56021927 | Pre-dose, and post-dose Day 1 (0.5, 1, 1.5, 2, 4, 6, 8, 12, 24 hours), Day 2, 3, 4, 5, 6, 7, 8, 15, 22, 29, 36, 43, 50, 57
  Relative bioavailability is the percentage of the administered dose that is systemically available.
Metabolite to Parent Drug Ratio for Cmax of JNJ-56021927 | Pre-dose, and post-dose Day 1 (0.5, 1, 1.5, 2, 4, 6, 8, 12, 24 hours), Day 2, 3, 4, 5, 6, 7, 8, 15, 22, 29, 36, 43, 50, 57
  Metabolite to parent drug ratio for maximum observed plasma concentration.
Metabolite to Parent Drug Ratio for AUClast of JNJ-56021927 | Pre-dose, and post-dose Day 1 (0.5, 1, 1.5, 2, 4, 6, 8, 12, 24 hours), Day 2, 3, 4, 5, 6, 7, 8, 15, 22, 29, 36, 43, 50, 57
  Metabolite to parent drug ratio for area under the plasma concentration time curve from time 0 to time of the last observed quantifiable concentration (Clast).
Metabolite to Parent Drug Ratio for AUCinfinity of JNJ-56021927 | Pre-dose, and post-dose Day 1 (0.5, 1, 1.5, 2, 4, 6, 8, 12, 24 hours), Day 2, 3, 4, 5, 6, 7, 8, 15, 22, 29, 36, 43, 50, 57
  Metabolite to parent drug ratio for area under the plasma concentration time curve from time 0 to infinite time, calculated as the sum of AUClast and Clast/ first-order rate constant, in which Clast is the last observed quantifiable concentration.
Number of Participants With Adverse Events as a Measure of Safety and Tolerabilty | Up to Day 57

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Tempe, Arizona, United States